CLINICAL TRIAL: NCT00845468
Title: Coronary Flow Velocity Reserve According to Glucometabolic State in Acute Myocardial Infarction; Relation to Ventricular Systolic and Diastolic Function
Brief Title: Coronary Flow Reserve and Glucometabolic State
Status: Completed | Type: Observational
Sponsor: Medicinsk Forsknings Afdeling (Other)
Responsible Party: Brian Bridal Løgstrup, Medicinsk Forskning Afdeling
Other Study IDs: 07-4-B368-A1392-22379; VF 20050103
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Acute Myocardial Infarction; Diabetes Mellitus; Prediabetes
Keywords: coronary flow reserve; diabetes mellitus; acute myocardial infarction; transthoracic echocardiography
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
Diabetes mellitus is a major risk factor for the development of ischemic heart disease, and patients with diabetes mellitus have a worse outcome following an acute myocardial infarction than non-diabetic patients. Furthermore, abnormal glucose metabolism below the diagnostic threshold of diabetes mellitus is also associated with increased risk of death compared to patients with a normal glucose metabolism. The frequency of abnormal glucose metabolism in acute myocardial infarction is high, and approximately 70% of myocardial infarction patients have diabetes mellitus, newly diagnosed diabetes mellitus or impaired glucose tolerance, leaving only 30% with normal glucose metabolism. The increased mortality among patients with acute myocardial infarction and abnormal glucose metabolism seems mainly related to a higher occurrence of congestive heart failure, suggesting that an abnormal glucose metabolism may play an important role among others in endothelial dysfunction, infarct healing and overall left ventricle function. This raises the question, whether patients with acute myocardial infarction and abnormal glucose metabolism have increased frequency of micro- or macrovascular disease or both.

Coronary flow velocity reserve reflects the patency of the epicardial coronary artery in combination with vasodilator capacity of the microcirculation and may therefore offer a tool for assessment of macro- and microcirculation.

This study will focus on the relation between coronary flow velocity reserve estimated by transthoracal Doppler echocardiography and mortality, risk for heart failure and left ventricle function after acute myocardial infarction stratified according to glycometabolic state

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed first AMI based on characteristic clinical symptoms and/or electrocardiographic signs of AMI and Troponin T or I or CK-MB over diagnostic limits for AMI
2. Referral for coronary arteriography based on the actual myocardial infarction
3. Written informed consent

Exclusion Criteria:

1. Previous myocardial infarction
2. Asthma bronchiale
3. 2 or/and 3 degree atrio-ventricular block and paced rhythm
4. Mental state that makes the patient unavailable in attending the study
5. Use of dipyridamol
6. Sick Sinus Syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from a acute myocardial infarction
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian B Løgstrup, MD, Principal Investigator — Medicinsk Forsknings Afdeling
Locations (1):
- Hospital of Fünen Svendborg, Svendborg, Svendborg, Denmark

REFERENCES:
- [Derived] Logstrup BB, Hofsten DE, Christophersen TB, Moller JE, Botker HE, Pellikka PA, Egstrup K. Influence of abnormal glucose metabolism on coronary microvascular function after a recent myocardial infarction. JACC Cardiovasc Imaging. 2009 Oct;2(10):1159-66. doi: 10.1016/j.jcmg.2009.06.012. PMID 19833304